CLINICAL TRIAL: NCT01410383
Title: A Placebo-controlled, Double-blind, Randomised, Parallel-group, Long Term Phase III Trial Assessing the Safety and Efficacy of Eprotirome in Patients With Heterozygous Familial Hypercholesterolaemia Who Are on Optimal Standard of Care
Brief Title: Efficacy and Safety Study of Eprotirome in HeFH Patients Who Are on Optimal Standard of Care
Acronym: AKKA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Karo Bio AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KBT 009
Record Dates: First submitted 2011-07-13; First posted 2011-08-05 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Heterozygous Familial Hypercholesterolaemia
Keywords: hypercholesterolemia,; dyslipidemia,; thyroid,; safety,; Heterozygous Familial Hypercholesterolaemia; coronary artery disease
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias; Thyroid Diseases; Coronary Artery Disease | interventions — 3-((3,5-dibromo-4-(4-hydroxy-3-(1-methylethyl)phenoxy)phenyl)amino)-3-oxopropanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Eprotirome I (Experimental)
  Interventions: Drug: Eprotirome
- Eprotirome II (Experimental)
  Interventions: Drug: Eprotirome

INTERVENTIONS:
Drug: Placebo — Tablets taken daily
  Arms: Placebo
Drug: Eprotirome — Tablets taken daily
  Other Names: KB2115
  Arms: Eprotirome I
Drug: Eprotirome — Tablets taken daily
  Other Names: KB2115
  Arms: Eprotirome II

SUMMARY:
Eprotirome is a liver selective thyroid hormone that can reduce several independent risk factors for cardiovascular disease, while an euthyroid state is preserved in the extrahepatic tissue.

The purpose of this Phase III study is to assess the long-term efficacy and safety of Eprotirome in Patients with heterozygous Familial Hypercholesterolaemia who are on optimal standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed HeFH and 18 years of age at screening
* Presence of clinical atherosclerotic disease that confers high risk for CAD events together with an LDL-C more than 2 mmol/L (more than 80 mg/dL)
* Presence of risk factors for CVD (other than the HeFH diagnosis) together with an LDL-C more than 2.5 mmol/L (more than 100 mg/dL)
* On an optimal standard of care, defined as being on a stable dose of statin (rosuvastatin, atorvastatin, or simvastatin) with or without ezetimibe for 8 weeks prior to randomisation

Exclusion Criteria:

* Significant health problems in recent past including heart failure,cardiac electrophysiologic instability, rheumatoid arthritis, thyroid dysfunction, liver disease, cancer, secondary dyslipidaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Percent reduction in low-density lipoprotein cholesterol (LDL-C) from baseline | 12 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Kastelein, Professor, Principal Investigator — Academic Medical Center (AMC) of the University of Amsterdam

REFERENCES:
- [Derived] Sjouke B, Langslet G, Ceska R, Nicholls SJ, Nissen SE, Ohlander M, Ladenson PW, Olsson AG, Hovingh GK, Kastelein JJ. Eprotirome in patients with familial hypercholesterolaemia (the AKKA trial): a randomised, double-blind, placebo-controlled phase 3 study. Lancet Diabetes Endocrinol. 2014 Jun;2(6):455-63. doi: 10.1016/S2213-8587(14)70006-3. Epub 2014 Feb 18. PMID 24731671